CLINICAL TRIAL: NCT03344406
Title: Assessing the Adequacy of the Evaluating Respiratory Symptoms in COPD (E-RS:COPD™) Measure Among Patients With Moderate to Severe Asthma
Brief Title: A Study to Evaluate Conceptual Saturation of Evaluating Respiratory Symptoms (E-RS) in Subjects With Asthma
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Evidera (Industry)
Responsible Party: Sponsor
Other Study IDs: 206605
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Asthma
Keywords: Asthma; Telephone interview; Cross-sectional; Qualitative research; E-RS: COPD
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with asthma: Subjects with moderate to severe asthma will be interviewed via telephone. Subjects will complete a daily diary including the E-RS: COPD and supplemental asthma items for 7 days.
  Interventions: Other: Telephonic interviews; Other: E-RS: COPD; Other: Supplemental asthma items; Other: Daily diary; Other: Sociodemographic questionnaire; Other: Clinical questionnaire

INTERVENTIONS:
Other: Telephonic interviews — Qualitative concept elicitation telephone interviews will be conducted in subjects with asthma.
Other: E-RS: COPD — E-RS questionnaire will directly measure respiratory symptom severity.
Other: Supplemental asthma items — Supplemental asthma items will include one question on wheeze and an item on breathlessness with activities to evaluate shortness of breath associated with strenuous activities.
Other: Daily diary — Subjects will complete a daily diary including the E-RS: COPD and supplemental asthma items for 7 days.
Other: Sociodemographic questionnaire — Sociodemographic questionnaire will capture subject's demographic characteristics, including age, gender, and the highest level of educational attainment.
Other: Clinical questionnaire — Clinical questionnaire will capture subject's clinical characteristics including the number of asthma exacerbations in the past 12 months, absenteeism due to asthma in the past month, and the presence of comorbid conditions.

SUMMARY:
Asthma and chronic obstructive pulmonary disease (COPD) are chronic inflammatory conditions involving the small airways with airflow limitations resulting from genetic and environmental interactions. Currently, there are no existing subject diaries with evidence of responsiveness to measure the daily symptoms of asthma. Therefore, there is a need to either develop a new symptom diary to characterize subject burden of asthma symptoms or modify/adapt an existing tool from a related disease area for use in subjects with moderate to severe asthma. The E-RS in COPD (E-RS: COPD®) questionnaire was developed as a measure of daily respiratory symptoms associated with COPD. The fixed dose combination of fluticasone furoate/ umeclidinium/ vilanterol (FF/UMEC/VI) administered via the ELLIPTA® dry powder inhaler (DPI) has been developed for the treatment of asthma. This cross-sectional, qualitative study is designed to understand the symptoms and disease experience of subjects with moderate to severe asthma. This study will also evaluate underlying concepts that are most important to asthmatic subjects compared to symptoms and concepts included in the E-RS: COPD and two supplemental asthma items (wheeze and shortness of breath with physical activity). Approximately 32 subjects will be included in the study and interviewed via telephone. Each interview including time for consent, qualitative interview, and completion of case report forms (CRFs) is expected to last approximately 60 to 90 minutes. Subjects will be expected to complete a daily diary for the next 7 days, following the initial telephone interview. E-RS: COPD and ELLIPTA are registered trademarks of GlaxoSmithKline group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older at the time of consent.
* History of airflow obstruction as indicated by a pre-bronchodilator forced expiratory volume in one second (FEV1) <80 percent predicted recorded in the previous 12 months.
* Documented evidence of a reversibility assessment within the previous 12 months, which demonstrated a post-bronchodilator increase in FEV1 of >=12 percent and >= 200 milliliters (mL).
* Diagnosed with moderate or severe asthma as defined by a stable maintenance inhaled corticosteroid (ICS) dose for at least 12 weeks prior to screening of; moderate: medium ICS dose > 250 and <=500 micrograms per day (mcg/day) fluticasone propionate (or equivalent) based on the total daily maintenance treatment dose; Severe: high ICS dose > 500 mcg/day fluticasone propionate (or equivalent) based on the total daily maintenance treatment dose.
* Documented control status defined using the asthma control questionnaire (ACQ-6) items (ACQ-6) obtained at the time of screening.
* Able to understand, read and speak English or Spanish sufficiently to complete all assessments.
* Willing and able to take part in a telephone interview session.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Is a current smoker.
* Has any medical condition that would preclude participation in this study, including the presence of emphysema or chronic bronchitis (COPD other than asthma) or a clinically important lung condition other than asthma such as current infection, bronchiectasis, pulmonary fibrosis, bronchopulmonary aspergillosis or diagnoses of an eosinophilic disorder such as eosinophilic esophagitis or a history of lung cancer.
* Participated in an interventional study within the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 32 subjects with moderate to severe asthma will be included in the study. Of these, approximately 25 will be English-speaking and 5-7 Spanish-speaking subjects. All subjects will be recruited from up to approximately 10 clinical sites in the United States and Canada.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Number of subjects attending semi-structured interview | Up to 7 days
  A semi-structured interview guide will introduce and direct the discussion during the interview session. It will be used to elicit concepts of moderate to severe asthma symptoms and impacts as well as to assess the overall comprehension of the E-RS: COPD and supplemental asthma items. The interview guide is also designed to elicit from subjects how they used the provided response options to answer each item and provide them the opportunity to report if there are missing categories or if they could not respond to the item with the given response option.
Number of subjects completing E-RS questionnaire in COPD | Up to 7 days
  The E-RS: COPD questionnaire consists of 11 items from the 14 item exacerbations of COPD (EXACT-PRO) instrument. The 11-items will be scored on a 5-point scale ranging from "not at all" to "extreme". Items of the E-RS: COPD will capture information related to respiratory symptoms such as breathlessness, cough, sputum production, chest congestion, and chest tightness. The daily recording of information with the E-RS: COPD will allow assessment of underlying day-to-day variability of a subject's symptoms.
Number of subjects completing supplemental asthma items | Up to 7 days
  Two supplemental asthma items will be asked in conjunction with the E-RS: COPD questionnaire, including: a question on wheezing, a symptom of importance in asthma, and an item on breathlessness with activities to evaluate shortness of breath associated with strenuous activities.
Number of subjects completing daily diary | Up to 7 days
  Subjects will complete a paper-pen daily diary including the E-RS: COPD and supplemental asthma items for 7 days. Several questions related to the relevance of the E-RS: COPD and supplemental asthma items will be asked to subjects.
Number of subjects completing sociodemographic questionnaire | Up to 7 days
  The sociodemographic questionnaire is a brief, self-administered questionnaire, which includes items to capture subject's demographic characteristics, including age, gender, and the highest level of educational attainment. Subjects will complete the sociodemographic questionnaire at the time of the interview.
Number of subjects completing clinical questionnaire | Up to 7 days
  The clinical questionnaire is a brief, self-administered questionnaire, which includes questions about the number of asthma exacerbations in the past 12 months, absenteeism due to asthma in the past month, and the presence of comorbid conditions. Subjects will complete the clinical questionnaire at the time of the interview.
Time to diagnosis of asthma based on clinical data form | Up to 7 days
  Clinicians will complete time to asthma diagnosis in clinical data form for each subject upon enrollment.
Number of subjects with exacerbation history based on clinical data form | Up to 7 days
  Clinicians will complete exacerbation history in clinical data form for each subject upon enrollment.
Number of subjects with other health conditions based on clinical data form | Up to 7 days
  Clinicians will complete information of any other health condition in clinical data form for each asthmatic subject upon enrollment.
Number of subjects receiving maintenance therapy based on clinical data form | Up to 7 days
  Clinicians will complete information of subjects receiving maintenance therapy in clinical data form.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Pittsburgh, Pennsylvania, United States